

## PROTOCOL SUMMARY

TITLE: A Post-Market Study of Transcatheter Perivascular Renal

Denervation for the Treatment of Hypertension using the Ablative Solutions Inc. Peregrine System<sup>TM</sup> Infusion Catheter

**SHORT TITLE:** The Peregrine Post-Market Study

PROTOCOL ID: CR0001

INVESTIGATIONAL

**PRODUCT:** 

Peregrine System<sup>TM</sup> Infusion Catheter

**INDICATION:** Hypertension

ClinicalTrials.gov ID: NCT02570113

**PHASE:** Post market clinical follow up study

**SPONSOR:** Ablative Solutions, Inc.

6203 San Ignacio Avenue, Suite 110

San Jose, CA 95119, US

COORDINATING

**INVESTIGATORS:** 

Prof. Dr. med. Horst Sievert

**PROTOCOL VERSION:** Rev K

**DATE:** 16 April 2018

\*




| INVESTIGATIONAL PRODUCT | |
|---|---|
| Name of Product | Peregrine System <sup>TM</sup> Infusion Catheter |
| CLINICAL CONDITION/IND | ICATION |
| Hypertension | |
| Protocol ID | CR0001 |
| Protocol Title | A Post-Market Study of Transcatheter Perivascular Renal Denervation for the Treatment of Hypertension using the Ablative Solutions Inc. Peregrine System <sup>TM</sup> Infusion Catheter |
| Short Title | The Peregrine Post-Market Study |
| Study Phase | Post market clinical follow up study |
| PLANNED STUDY PERIOD | |
| Initiation | November 2015 |
| <b>Study Completion</b> | May 2019 |
| Duration | Approximately 3.5 years |
| STUDY OBJECTIVES AND P | URPOSE |

## **Study Purpose**

To collect additional safety and performance data pertaining to renal denervation by using dehydrated alcohol as a chemical neurolytic agent delivered into the adventitial/peri-adventitial area of the renal arteries for the purpose of renal denervation, using the Peregrine Catheter, in patients with hypertension.

## **Objective**

The objectives of this post-market study are to collect additional safety and performance data pertaining to renal denervation by using dehydrated alcohol as a chemical neurolytic agent delivered into the adventitial/peri-adventitial area of the renal arteries for the purpose of renal denervation, using the Peregrine Catheter, in patients with hypertension.

| STUDY DESIGN | |
|---|---|
| Study Type/ Classification/<br>Discipline | Post market clinical follow up study for safety and performance (ambulatory blood pressure monitoring [ABPM], office blood pressure) |
| <b>Study Indication Type</b> | Treatment |




| Study Design | This post-market study is a prospective, single arm, open label, multicenter trial. Up to 60 subjects with hypertension will be treated with 0.6 mL of dehydrated alcohol as the neurolytic agent per renal artery. The data of the first 5 treated subjects in the study (including renal duplex ultrasound) will be assessed at the 1-month follow-up by the Data Safety Monitoring Board (DSMB). If no safety concern arises, treatment with 0.6 mL of alcohol will continue according to the protocol. Contenting subjects will be assessed for eligibility and baseline data collected. Subjects will attend the study site for the day of procedure. Subjects will be discharged from the study site per the physician's judgment. Subjects must be maintained on his/her baseline anti-hypertensive medications at the same doses through the 6 months follow up visit unless the study subject has symptomatic hypotension requiring anti-hypertensive medication reduction. Planned increases in anti-hypertensive medications must be in alignment with JNC-8 and/or European Hypertension Guidelines and with approval from the sponsor. |
|---|---|
| | months post-procedure. |
| Study<br>Geography/<br>Number of<br>Planned<br>Investigational<br>Sites | Europe: up to 10 sites in Europe. |
| Number of<br>Groups/ Arms/<br>Cohorts | 1 group |
| Number of<br>Subjects | Up to 60 |
| Planned Duration of Subject Participation | Up to 12 months |
| INVESTIGATIO | INVESTIGATIONAL PRODUCT |
| Product | Peregrine System <sup>TM</sup> Infusion Catheter used to deliver a neurolytic agent (such as dehydrated alcohol) to the perivascular area of the renal arteries to ablate the afferent and efferent sympathetic nerves serving the kidneys Dose: 0.6 mL alcohol per treated renal artery. Mode of administration: Direct infusion to the perivascular space, during an endovascular procedure |
| - | ction rolled in the study at the time they sign the informed consent form. No study-specific performed until after the subject has provided written informed consent. |


procedures will be performed until after the subject has provided written informed consent.



# **Subject Inclusion Criteria**

Subjects must meet ALL of the following inclusion criteria to receive the percutaneous procedure:

- 1. Adult subject, age 18-80, male or female
- 2. Subject has a target treatment vasculature diameter of  $\geq$ 4 mm and  $\leq$  7 mm and length of  $\geq$ 5 mm
- 3. Subject has 3 measurements with a mean of office Systolic Blood Pressure of ≥150 mmHg AND office Diastolic Blood Pressure of ≥85 mmHg
- 4. Subject has a 24-hour mean systolic Ambulatory Blood Pressure Measurement (ABPM) ≥135 mm Hg with ≥70% valid readings (as determined by measurement device)
- 5. Subject with hypertension is receiving and adhering to a stable medication regimen of at least 3 anti-hypertensive medications of different classes (for at least 4 consecutive weeks), one of which must be a diuretic
- 6. Subject agrees to have all study procedures performed, to comply with medication regimen and is able and willing to comply with all study follow-up visits
- 7. Subject has provided written informed consent

### **Exclusion Criteria**

Any subject who meets ANY of the following exclusion criteria will not receive the percutaneous interventional procedure:

- 1. Subject has a contraindication known for conventional percutaneous interventional procedures such as:
  - intolerance for antiplatelet/anticoagulant therapy
  - known allergy to contrast media
  - bleeding disorders (such as bleeding diathesis, thrombocytopenia and severe anemia)
- 2. Subject has documented severe untreated obstructive sleep apnea (Apnea Hypopnea Index [AHI] ≥30 per hour)
- 3. Subjects with nephrotic syndrome
- 4. Subjects on immunosuppressive medications or immunosuppressive doses of steroids
- 5. Subject has type 1 diabetes mellitus
- 6. Subject is pregnant or nursing or planning to become pregnant
- 7. Subject has an estimated glomerular filtration rate (eGFR) ≤20 mL/min/1.73m², based on the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation
- 8. Subject has imaging-assessed renal artery anatomy abnormalities or variations based on Investigator's evaluation of the screening images [i.e. magnetic resonance angiogram/angiography (MRA)/ computed tomography angiogram/angiography (CTA) examination and/or renal angiography]) meeting one of the following criteria:
  - Renal artery stenosis >60% of the normal diameter segment (diameter stenosis, compared to the angiographically normal proximal or distal segment)




- Any renal artery abnormality or disease that, per the physician assessment, precludes the safe insertion of the guiding catheter (such as but not limited to severe renal artery aneurysm, excessive tortuosity, severe renal artery calcification)
- Previous renal angioplasty associated with stenting or other implants, that, per the physician's
  assessment, precludes the safe deployment of the Peregrine catheter components in the target
  treatment segment of the renal artery
- 9. Subject has a history of nephrectomy, a single kidney or kidney tumor, or urinary tract obstruction (with potential for hydronephrosis)
- 10. Subject is known to have a non-functioning kidney or unequal renal size (>2 cm difference in renal length between kidneys associated with a chronic kidney disease or a deterioration of the kidney function)
- 11. Subject has a renal transplant
- 12. Subject has a history of myocardial infarction, unstable angina pectoris, or stroke/transient ischemic attack (TIA) within the last six months from planned procedure
- 13. Subject has hemodynamically significant valvular heart disease
- 14. Subject has heart failure (New York Heart Association [NYHA] III or IV) or has an ejection fraction ≤30%
- 15. Subject with chronic atrial fibrillation
- 16. Subjects who are allergic or intolerant of the neurolytic agent (such as dehydrated alcohol)
- 17. Any contraindication to the imaging as required per the protocol
- 18. Subject has a life expectancy of <12 months
- 19. Subject is currently enrolled in other potentially confounding research, i.e., another therapeutic or interventional research trial. Subjects enrolled in observational registries may still be eligible

